CLINICAL TRIAL: NCT00741572
Title: Individual Sensitivity for Interstitial Lung Diseases
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Dr. A.W. Boots, Maastricht University
Other Study IDs: MEC 08.3.048
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2009-09

CONDITIONS: Interstitial Lung Diseases
Keywords: sarcoidosis; fibrosis; oxidative stress; inflammation; triggers; individual sensitivity
MeSH Terms: conditions — Lung Diseases, Interstitial; Sarcoidosis; Fibrosis; Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The patients will be asked to donate 5L exhaled air and 20 ml blood.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
Interstitial lung diseases (ILD) is a collective noun for various chronic lung diseases, including sarcoidosis and idiopathic lung fibrosis (IPF). Sarcoidosis is a multi-systemic disease that includes damage to the lungs in 90% of the patients. Generally, the disease can be described as a systemic, granulomatous and antigen-driven disorder. IPF is a disease of only the lungs, in which an unknown cause induces a strong inflammation reaction leading to acute lung damage that ultimately results in the formation of scar tissue and stiffness of the lungs.

Unfortunately, the exact cause of ILD is still unknown. It is suggested that environmental and work-related exposure to various triggers can exert an effect on the course of the diseases. Examples of such triggers include bacteria, organic agents such as pollen and cotton dust and inorganic agents like metals and talc. Due to this unknown cause, it is difficult to treat ILD. Consequently, the current guideline is no medication or anti-inflammatory agents in severe cases. Unfortunately, this therapy is not completely effective.

Triggers that are suggested to cause ILD can exert their effects via various mechanisms. On the one hand, they can induce an inflammatory reaction as we recently demonstrated for various triggers including instillation material and sicila. During such an inflammatory reaction, cytokines are released that can induce oxidative stress, i.e. an imbalance between the formation of and the protection against reactive oxygen species (ROS). On the other hand, ILD-inducing triggers may directly cause an increased ROS production that subsequently can evoke an inflammatory reaction.

The objective of the current study is to investigate the individual sensitivity for the development of ILD after exposure to various triggers. Main focus will be the differences in the formation of and the protection against ROS as well as the occurring inflammatory reaction after exposure to such triggers.

Furthermore, a simple blood test will be developed to study and eventually even predict the individual reaction of subjects to various triggers.

Finally, to fully characterize the development of ILD after exposure to various triggers, the exhaled air of patients will be studied in order to identify specific markers of oxidative stress and damage.

ELIGIBILITY:
Inclusion Criteria:

* ILD diagnosis confirmed by lung biopsy, X ray or BALF analysis

Exclusion Criteria:

* smoking
* pregnancy or lactation
* use of vitamins or nutritional supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in this study include both men and women, who are 18 years of age or older and diagnosed with ILD using lung biopsy, X ray or BALF (broncho-alveolar lavage fluid) analysis and are either treated for this with anti-inflammatory agents or not. There's no maximum age set for this study since ILD can occur at all ages. Additional criteria are non smoking, no pregnancy or lactation and no use of vitamins or nutritional supplements.
  The inclusion of both treated and untreated patients enables us to study the effectiveness of anti-inflammatory agents on a larger scale.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
differences in the production of and the protection against ROS | 6 hours
differences in the occurring inflammatory reaction | 6 hours

SECONDARY OUTCOMES:
differences in the presence of so-called volatile organic compounds (VOCs) in the exhaled air | 0 hour

CONTACTS AND LOCATIONS:
Overall Officials: Aalt Bast, PhD, Study Chair — Maastricht University; Marjolein Drent, PhD, MD, Study Director — Maastricht University Medical Center; Agnes W Boots, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands

REFERENCES:
- [Derived] Fijten RRR, Smolinska A, Drent M, Dallinga JW, Mostard R, Pachen DM, van Schooten FJ, Boots AW. The necessity of external validation in exhaled breath research: a case study of sarcoidosis. J Breath Res. 2017 Nov 29;12(1):016004. doi: 10.1088/1752-7163/aa8409. PMID 28775245